CLINICAL TRIAL: NCT06028971
Title: Safety and Performance of the Biphasic Plate Distal Femur: A Multicenter Case Series
Status: Active, not recruiting | Type: Observational
Sponsor: 41medical AG (Industry)
Collaborators: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1156
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Distal Femur Fracture; Periprosthetic Fractures; Intra-Articular Fractures; Supracondylar Fracture
Keywords: Biphasic Plate DF; Distal Femur Fracture; Femur Fracture; Periprosthetic Fractures; Intra-Articular Fractures
MeSH Terms: conditions — Femoral Fractures, Distal; Periprosthetic Fractures; Intra-Articular Fractures; Femoral Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational multicenter case series is to assess the safety and performance of the CE-marked "Biphasic Plate Distal Femur" during standard of care.

DETAILED DESCRIPTION:
The goal of this observational study is to assess the safety and performance of the CE-marked "Biphasic Plate Distal Femur" during standard of care. The study is conducted as a retrospective and prospective multicenter case series. Eligible patients are those with fractures of the distal femur who are treated with the Biphasic Plate DF according to the Instruction for Use (IFU). The patient will be followed-up until healing or up to 12 months, whichever comes first.

To assess the safety and performance following data is collected:

* incidents of AEs/SAEs occurring in the affected lower extremity/extremities
* Bone healing assessed by a surgeon
* Weightbearing and function
* Patients' quality of life and pain level

ELIGIBILITY:
Inclusion Criteria:

* Patients with fractures of the distal femur requiring internal fixation and treated with the Biphasic Plate DF as indicated according to the IFU. As per the IFU, the Biphasic Plate DF is indicated for:

  * Distal shaft fractures
  * Supracondylar fractures
  * Intraarticular fractures
  * Periprosthetic fractures
* No other major implant beside the Biphasic Plate DF is used for fixation of the distal femur fracture, with the exceptions of lag screw(s) and/or cerclage wire(s), and/or a joint replacement.
* Patients who are willing and able to comply with postoperative FUs per local standard of care.
* Ability to provide informed consent according to the IRB/EC defined and approved procedures.
* Patients over 18 years of age

Exclusion Criteria (preoperatively):

* Patient is participating in another interventional clinical trial.

Exclusion Criteria (intraoperatively):

* Change of surgical plan intraoperatively at the discretion of the surgeon that Biphasic Plate DF is not used
* Necessity to apply a second (medial) plate (double plating) or an intramedullary nail in case of critical fixation distally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eledgible patients will be identified at the sites (primary care clinics)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of AEs/SAEs in the affected lower extremity/extremities | until clinically healed or up to 12 months
  The primary outcome measure is the occurrence of AEs/SAEs in the affected lower extremity/extremities that are deemed related, probably related, or possibly related to the surgical procedure or the Biphasic Plate DF

SECONDARY OUTCOMES:
Bone Healing | until clinically healed or up to 12 months
  Radiographic bone healing assessment using the modified Radiographic Union Scale for Tibia (mRUST) Score (1: Callus absent, visible fracture line, 2: Callus present, visible fracture line, 3: Callus bridging, visible fracture line, 4: Callus remodeled, invisible fracture line)
  Bone healing as assessed by the surgeon
Patient-reported outcome measures | until clinically healed or up to 12 months
  Quality of life questionaire Pain NRS (0-10) upon weightbearing

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Sommer, Dr. med., Principal Investigator — Kantonsspital Graubünden Chur
Locations (5):
- Germany (2):
  - Univeritätsklinikum Münster, Münster, North Rhine-Westphalia
  - Diakonie Jung-Stilling Siegen, Siegen, North Rhine-Westphalia
- Switzerland (3):
  - Universitätsspital Zürich, Zurich, Canton of Zurich
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
  - Universitätsspital Basel, Basel

IPD SHARING:
Plan to Share IPD: No